CLINICAL TRIAL: NCT04618900
Title: Osteotome-mediated Sinus Floor Elevation With Bio-Oss Collagen Compared With the Use of no Grafting Material. A Randomized Controlled Trial
Brief Title: Osteotome-mediated Sinus Floor Elevation With or Without Grafting Material
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Thomas Starch-Jensen, Professor, DDS, PhD, Aalborg University Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Aalborg University Hospital
Record Dates: First submitted 2020-11-02; First posted 2020-11-06 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Survival, Prosthesis; Bone Loss; Patient Satisfaction
Keywords: Alveolar ridge augmentation; Maxillary sinus floor elevation; Bone substitute
MeSH Terms: conditions — Prosthesis Failure; Bone Diseases, Metabolic; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant
Masking Description: Healthy patients in need of dental implant in the posterior part of the maxilla
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Osteotome-mediated sinus floor elevation with Bio-Oss collagen (Experimental): Sinus floor elevation with a grafting material (Bio-Oss collagen)
  Interventions: Procedure: Sinus floor elevation with a grafting material
- Osteotome-mediated sinus floor elevation with no grafting material (Placebo Comparator): Sinus floor elevation with no grafting material
  Interventions: Procedure: Sinus floor elevation with a grafting material

INTERVENTIONS:
Procedure: Sinus floor elevation with a grafting material — The use of grafting material for sinus floor elevation

SUMMARY:
Implant placement in the posterior part of the maxilla is frequently compromised or impossible due to atrophy of the alveolar process and pneumatisation of the maxillary sinus. Therefore, alveolar ridge augmentation is frequently necessary before or in conjunction with implant placement. The most commonly used method to augment the maxillary premolar and molar region involves the maxillary sinus floor augmentation applying the lateral window technique with a grafting material. However, the lateral window technique is associated with prolonged patient treatment time and increased morbidity. Thus, osteotome-mediated sinus floor elevation (OSFE) with or without the use of a grafting material has been advocated, when the residual bone height is more than 6 mm.

OSFE involves preparation of implant site through the use of concave osteotomes and elevation of the maxillary sinus floor. The survival of suprastructure and implants after OSFE with or without the use of a grafting material has never been assessed in long-term randomized controlled trials. A long-term study concluded that OSFE with no grafting material is a predictable treatment modality. High short-term implant survival rates after OSFE with or without the use of a grafting material have been reported in systematic reviews. However, the amount of new bone formation after OSFE with the use of a grafting material is significantly higher compared to the use of no grafting material, as documented in a systematic review. Harvesting of autogenous bone graft is associated with risk of donor site morbidity and bone substitutes of natural transplants involves a risk of contamination, activation of host immune system and disease transmission as well as they can be refused by patients for religious reasons or because they are in contrast with chosen lifestyle.

Therefore, the objective of the present study is to test the H0-hypothesis of no difference in the long-term implant treatment outcome after OSFE with Bio-Oss Collagen compared with the use of no grafting material. A total of 40 consecutively healthy patients with a missing posterior tooth in the maxilla will be allocated at random to OSFE with Bio-Oss Collagen or no grafting material and simultaneous implant placement. Clinical and/or radiographical evaluation using periapical radiographs and Cone Beam Computer Tomography (CBCT) will be performed preoperatively, immediate postoperatively, after abutment connection, after prosthetic rehabilitation, one year, three years and five years after loading to assess the long-term implant treatment outcome and the volumetric changes of the augmented area. The primary outcome will include survival of suprastructures, survival of implants, volumetric stability of the augmented area, peri-implant marginal bone level, oral health related quality of life, and complications related to the two treatment modalities.

DETAILED DESCRIPTION:
Implant placement in the posterior part of the maxilla is frequently compromised or impossible due to atrophy of the alveolar process and pneumatisation of the maxillary sinus. Therefore, alveolar ridge augmentation is frequently necessary before or in conjunction with implant placement. The most commonly used method to augment the maxillary premolar and molar region involves the maxillary sinus floor augmentation applying the lateral window technique with autogenous bone graft or bone substitutes and the treatment outcome has been reported in systematic reviews. However, maxillary sinus floor augmentation with the lateral window technique and bone harvesting is associated with prolonged patient treatment time and risk of donor site morbidity. Hence, OSFE with or without the use of a grafting material is commonly used to simplify the surgical procedure, when the residual alveolar bone height is more than 6 mm.

OSFE with simultaneous implant placement was originally described by Summers in 1994. The surgical procedure involves a transalveolar up-fracture and elevation of the maxillary sinus floor and Schneiderian membrane using concave osteotomes. Implants are inserted simultaneously to support the elevated floor of the maxillary sinus. The created compartment between the elevated floor of the maxillary sinus and the original sinus floor is filled with either particulated autogenous bone graft, a bone substitute or without a grafting material. The final implant treatment outcome after OSFE with or without the use of a grafting material have previous been assessed in systematic reviews and meta-analyses disclosing high implant survival rates with few complications. However, the included studies are often characterized by a moderate to high risk of bias and the conclusions are based on short-term non-randomized controlled trials, whereas long-term randomized controlled trials assessing OSFE with or without the use of a grafting material is sparse.

OSFE with autogenous bone graft or a bone substitute is considered the golden standard and the gain in alveolar bone height is enhanced with the use of a grafting material compared to the use of no grafting material. Bio-Oss (Geistlich Pharma AG, Wolhusen, Switzerland) is a deproteinized bone substitute of bovine bone origin and several studies have documented that Bio-Oss possesses important properties when used as a membrane-supporting material and as a scaffold for in-growth of host cells including biocompatibility and osteoconductivity. Bio-Oss has been used for different bone augmentation procedures for more than 30 years and OSFE with Bio-Oss is a safe and very predictable surgical procedure with few complications and minimal morbidity, as documented in systematic reviews and long-term studies. However, bone substitutes of natural transplants involves a risk of contamination, activation of host immune system and disease transmission as well as they can be refused by patients for religious reasons or because they are in contrast with chosen lifestyle. Thus, OSFE without a grafting material is associated with obvious advantages for the patient, including reduced risk of infection, less cost, reduced length of operation time and no risk of disease transmission.

Survival of suprastructures and implants are the most important measures for the assessment of the long-term implant treatment outcome. However, long-term survival of suprastructures after OSFE with or without the use of a grafting material has never been compared within a randomized controlled trial. Moreover, patient-reported outcome measures after OSFE have never previously been assessed. A long-term randomized controlled trial revealed no significant differences in implant survival after OSFE with Bio-Oss compared with the use of no grafting material after five years. A newly published systematic review and meta-analysis disclosed no significant differences in the short-term implant survival after OSFE with or without the use of a grafting material and a long-term retrospective study assessing OSFE without the use of a grafting material reported an implant survival rate 97.7% after 15 years. Moreover, long-term studies assessing OSFE without a graft material revealed high implant survival after 10 years.

In conclusion, OSFE without the use of a grafting material seems to be a predictable treatment modality with high implant survival. However, the long-term survival of suprastructure and implants after OSFE with or without the use of a graft material is presently not sufficient clarified and has not been assessed in long-term randomized trial.

ELIGIBILITY:
Inclusion Criteria:

* Male and females of ≥20 years of age.
* Missing one posterior maxillary tooth (premolar or molar) for more than 4 months.
* Residual vertical alveolar bone height of the maxillary alveolar process ≤ 6-10mm ≤.
* Width of the alveolar maxillary process ≥6.5 mm.
* Mandibular occluding teeth.
* Should be able to speak and understand Danish.

Exclusion Criteria:

* Medical contraindications to implant therapy e.g. recent myocardial infarction and cerebrovascular accident, recent valvular prosthesis surgery, immunosuppression, bleeding issues, active treatment of malignancy, drug abuse, psychiatric illness and intravenous bisphosphonate treatment.
* Irradiated jaw bones (radiotherapy treatment).
* Full mouth plaque score >25%.
* Progressive marginal periodontitis in the maxilla and mandible.
* Acute infection in the area intended for implant placement.
* Parafunction, bruxism, or clenching.
* Psychiatric problems or unrealistic expectations.
* Heavy tobacco use, define as >10 cigarettes per day.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-11-22 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Survival of suprastructures and implants | 1-year
  Loss of suprastructures and dental implants

SECONDARY OUTCOMES:
Volumetric stability of the grafting material | 1-year
  Radiographic loss of the augmented area

CONTACTS AND LOCATIONS:
Locations (1):
- Aalborg University Hospital, Aalborg, North Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared with other researchers

REFERENCES:
- [Derived] Starch-Jensen T, Bruun NH, Spin-Neto R. Endo-sinus bone gain following osteotome-mediated sinus floor elevation with Bio-Oss Collagen compared with no grafting material: a one-year single-blind randomized controlled trial. Int J Oral Maxillofac Surg. 2023 Nov;52(11):1205-1215. doi: 10.1016/j.ijom.2023.03.009. Epub 2023 Mar 29. PMID 36997448